CLINICAL TRIAL: NCT06115499
Title: Phase II/III Second-Line NABPLAGEM vs. Nab-Paclitaxel/Gemcitabine in BRCA1/2 or PALB2 Mutant Metastatic Pancreatic Ductal Adenocarcinoma (PLATINUM)
Brief Title: The PLATINUM Trial: Optimizing Chemotherapy for the Second-Line Treatment of Metastatic BRCA1/2 or PALB2-Associated Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A022106; NCI-2023-06547 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Acinar Cell Carcinoma; Pancreatic Adenocarcinoma; Pancreatic Adenosquamous Carcinoma; Pancreatic Carcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Squamous Cell Carcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine; Cisplatin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (nab-paclitaxel, gemcitabine, cisplatin) (Experimental): Patients receive nab-paclitaxel IV over 30-40 minutes, gemcitabine IV over 30-40 minutes, and cisplatin IV over 30-60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI or CT throughout the trial. Patients may optionally undergo blood sample collection at baseline and on study.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography; Procedure: Biospecimen Collection
- Arm II (nab-paclitaxel, gemcitabine) (Active Comparator): Patients receive nab-paclitaxel IV over 30-40 minutes and gemcitabine IV over 30-40 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI or CT throughout the trial. Patients may optionally undergo blood sample collection at baseline and on study.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Nab paclitaxel — Given IV
  Other Names: ABI-007; Abraxane; Albumin-bound Paclitaxel; Protein-bound Paclitaxel
Drug: Gemcitabine — Given IV
Drug: Cisplatin — Given IV
  Arms: Arm I (nab-paclitaxel, gemcitabine, cisplatin)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; CT Scan
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase II/III trial compares the effect of the 3-drug chemotherapy combination of nab-paclitaxel, gemcitabine, plus cisplatin versus the 2-drug chemotherapy combination of nab-paclitaxel plus gemcitabine for the treatment of patients with pancreatic cancer that has spread to other places in the body (metastatic) and a known genetic mutation in the BRCA1, BRCA2, or PALB2 gene.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and compare overall response rate (ORR) in patients with BRCA1/2 or PALB2 mutant pancreas cancer whose disease has progressed on front-line fluorouracil, irinotecan, leucovorin and oxaliplatin (FOLFIRINOX) treated with nab-paclitaxel, gemcitabine, and cisplatin (NABPLAGEM) = nab-paclitaxel, gemcitabine, and cisplatin (arm 1) versus nab-paclitaxel and gemcitabine (arm 2). (Phase II) II. To evaluate and compare overall survival (OS) time in patients with BRCA1/2 or PALB2 mutant whose disease has progressed on front-line FOLFIRINOX treated with 1) NABPLAGEM = nab-paclitaxel, gemcitabine, and cisplatin (arm 1) versus nab-paclitaxel and gemcitabine (arm 2). (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate and compare progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) criteria between 2 treatment arms.

II. To evaluate and compare duration of response (DoR) between 2 treatment arms.

III. To evaluate and compare CA19-9 response (defined as patients with a baseline CA19-9 >= 2x upper limit of normal (ULN) who demonstrate a minimum 25% decrease in CA19-9 at any time point) between 2 treatment arms.

IV. To evaluate and compare toxicity profile as assessed by treating clinicians between 2 treatment arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nab-paclitaxel intravenously (IV) over 30-40 minutes, gemcitabine IV over 30-40 minutes, and cisplatin IV over 30-60 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) or computed tomography (CT) throughout the trial. Patients may optionally undergo blood sample collection at baseline and on study.

ARM II: Patients receive nab-paclitaxel IV over 30-40 minutes and gemcitabine IV over 30-40 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI or CT throughout the trial. Patients may optionally undergo blood sample collection at baseline and on study.

After completion of study treatment, patients are followed up within 30 days and then every 3 months for 2 years or until death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic adenocarcinoma. Adenosquamous carcinoma, squamous carcinoma, acinar cell carcinoma, and carcinoma not otherwise specified are also acceptable
* BRCA1/2 or PALB2 mutation (somatic or germline) identified on any Clinical Laboratory Improvement Amendments (CLIA)-certified gene panel. Mutations must be considered pathogenic or likely pathogenic by a reference database such as ClinVar or OncoKb.org. (Submission of mutation report will be required)
* Measurable disease
* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment
* Clinical or radiographic progression on first-line FOLFIRINOX (or nanoliposomal irinotecan, fluorouracil, leucovorin, and oxaliplatin [NALIRIFOX]) for metastatic disease

  * Patients whose front-line chemotherapy was required to be simplified due to toxicity associated with any of the constituent components of FOLFIRINOX/NALIRIFOX (e.g. simplified to leucovorin calcium, fluorouracil, and oxaliplatin [FOLFOX], leucovorin calcium, fluorouracil, and irinotecan [FOLFIRI], fluorouracil [5-FU] [including capecitabine]) will be eligible
  * Patients with progressive disease while on maintenance PARP inhibitor treatment after FOLFIRINOX (or NALIRIFOX), irrespective of how long ago they received FOLFIRINOX/NALIRIFOX, will also be eligible
  * Patients who develop metastatic disease during or within 6 months after completing FOLFIRINOX/NALIRIFOX in either the locally advanced or adjuvant/neoadjuvant settings will be eligible
* Patients may not have received prior cisplatin for their pancreatic cancer in any setting

  * Note: Patients may have previously received gemcitabine +/- nab-paclitaxel for resectable (neoadjuvant/adjuvant) or locally advanced disease if (1) treatment was completed > 1 year ago and (2) in the opinion of the treating provider, re-treatment with gemcitabine/nab-paclitaxel is appropriate
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky performance status >= 60)
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 8.0 g/dL
* Creatinine =< 1.8 x institutional upper limit of normal (ULN) or calculated creatinine clearance (Calc. CrCl) > 40 mL/min
* Total bilirubin =< 2.0 x institutional ULN

  * Any elevated bilirubin should be asymptomatic at enrollment (except for participants with documented Gilbert's syndrome who may only be included if the total bilirubin =< 3 x ULN or direct bilirubin =< 1.5 x ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 3 x institutional ULN

  * AST/ALT of =< 5 x ULN if liver metastases are present
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
* Patients with > grade 2 peripheral sensory neuropathy are not eligible
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 8-weeks.

  * Patients with known, new or progressive brain metastases (active brain metastases) or leptomeningeal disease are ineligible
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load anytime within 6 months prior to registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Concomitant chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study
* Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-12-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (Phase II) | Up to 12 months
  Will be assessed by the proportion of patients who achieve complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) during the protocol treatment. Fisher's exact test will be conducted based on the first 32 patients in each arm who meet PP population criteria.
Overall Survival (OS) (Phase III) | From the date of randomization to the date of death due to all causes, assessed up to 5 years
  Will be conducted on modified intention-to-treat population. Stratified Cox model will be constructed to compare OS in the experimental arm to OS in the control arm.

SECONDARY OUTCOMES:
Progression-free survival | From the date of randomization to the date of first documented disease progression or death due to all causes, whichever occurs first, assessed up to 5 years
  Will be assessed per RECIST 1.1. Will be estimated, in each arm, using the method of Kaplan-Meier and compared by stratified Cox regression model.
Incidence of adverse events | Up to 30 days after the last dose of study treatment
  The maximum grade for each type of adverse events that are possibly, probably, or definitely related to study treatments will be recorded for each patient.

CONTACTS AND LOCATIONS:
Locations (345):
- United States (345):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCI Health Laguna Hills, Laguna Hills, California
  - Mercy Cancer Center, Merced, California
  - Providence Queen of The Valley, Napa, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Saint Joseph's Medical Center, Stockton, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Hickman Cancer Center, Adrian, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Saint Joseph's Crosslake Clinic, Crosslake, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Essentia Health - Saint Joseph's Pequot Lakes Clinic, Pequot Lakes, Minnesota
  - Essentia Health - Saint Joseph's Pine River Clinic, Pine River, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health - Saint Joseph's Staples Clinic, Staples, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Tamarack Health Hayward Medical Center, Hayward, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Memorial Hospital of Laramie County, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Undecided